CLINICAL TRIAL: NCT00502476
Title: Multicenter Evaluation of The Effectiveness of Source Control With Daily Chlorhexidine Skin Preparation in Reducing Nosocomial Infections Including MRSA and VRE
Brief Title: Multicenter Trial of Daily Chlorhexidine Bathing to Reduce Nosocomial Infections
Acronym: CBET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Sage Products, Inc. (Industry)
Other Study IDs: CI06-003
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Nosocomial Bacteremia; MRSA Colonization; MRSA Infection; VRE Colonization; VRE Infection
Keywords: MRSA; VRE; BSI
MeSH Terms: interventions — Baths

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bathing with Chlorhexidine Impregnated Washcloths

SUMMARY:
To determine if daily bathing with chlorhexidine impregnated washcloths will reduce the incidence of MRSA and VRE within an Intensive Care Unit (ICU) or ward setting.

DETAILED DESCRIPTION:
This is a cluster randomized, crossover-controlled trial with wards as the units of randomization. The trial will predominantly take place in ICU's but may include any acute care ward that has active surveillance for MRSA and or VRE in place (i.e., Bone Marrow transplant units, Oncology wards, etc.) Units will be randomly assigned to utilize two bathing routines in a random order. Each bathing routine will be utilized on all admitted patients to the unit for a six month study period for a total study duration of 12 months. The two bathing routines will include either the use of the Comfort® Bath Washcloth System (control) or the use of 2% Chlorhexidine Gluconate Cloth. Randomized units will either start with 2% Chlorhexidine Gluconate Cloth for six months and then switch to Comfort™ Bath Washcloth for the remaining six month period or the reverse order. Data collection will include all surveillance and clinical cultures for MRSA and or VRE and all bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to study units during the proposed study interval are eligible for inclusion in the study

Exclusion Criteria:

* Patients with known allergies to chlorhexidine gluconate or any other ingredients in the product
* Patients with burns that include a high percentage of disrupted body surface area
* Use in patients undergoing lumbar punctures or contact with the meninges
* Patients with large open skin wounds; and
* Children less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2007-08; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Climo, MD, Study Director — Hunter Holmes Mcguire Veteran Affairs Medical Center; Edward S Wong, MD, Principal Investigator — Hunter Holmes Mcguire Veteran Affairs Medical Center; Jane A Cecil, MD, Principal Investigator — Hunter Holmes Mcguire Veteran Affairs Medical Center; Kent Sepkowitz, MD, Principal Investigator — Weil Medical College of Cornell University; Trish M Perl, MD, MSc, Principal Investigator — Johns Hopkins University; Debbie Yokoe, MD, MPH, Principal Investigator — Harvard School of Medicine, Brigham and Women's Hospital; Maureen Bolon, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Dave K Warren, MD, Principal Investigator — Washington University School of Medicine; Loreen Herwaldt, MD, Principal Investigator — University of Iowa
Locations (7):
- United States (7):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Barnes Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hunter Holmes McGuire Veteran Affairs Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Climo MW, Yokoe DS, Warren DK, Perl TM, Bolon M, Herwaldt LA, Weinstein RA, Sepkowitz KA, Jernigan JA, Sanogo K, Wong ES. Effect of daily chlorhexidine bathing on hospital-acquired infection. N Engl J Med. 2013 Feb 7;368(6):533-42. doi: 10.1056/NEJMoa1113849. PMID 23388005